CLINICAL TRIAL: NCT00230620
Title: Molecular Studies on Hereditary Haemorrhagic Telangiectasia Families With Pulmonary Arteriovenous Malformations
Brief Title: Molecular Studies on Hereditary Haemorrhagic Telangiectasia Families
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS1
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with HHT and their families: No intervention - blood or saliva sample only

SUMMARY:
This study will examine genes involved in the vascular dysplasia Hereditary haemorrhagic telangiectasia i(HHT)

DETAILED DESCRIPTION:
Hereditary haemorrhagic telangiectasia (HHT) is a condition inherited as an autosomal dominant trait. Sequencing DNA from affected and unaffected family members allows us to identify disease-causal genes. Sequencing these genes allows us to identify what the precise DNA variants are which are causing disease, particularly if linked to functional assays in separate studies.

ELIGIBILITY:
Inclusion Criteria:

* Member of family affected by HHT

Exclusion Criteria:

* Unable or unwilling to provide informed consent for DNA sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hereditary haemorrhagic telangiectasia and their families
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1998-12 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom

REFERENCES:
- [Result] Cole SG, Begbie ME, Wallace GM, Shovlin CL. A new locus for hereditary haemorrhagic telangiectasia (HHT3) maps to chromosome 5. J Med Genet. 2005 Jul;42(7):577-82. doi: 10.1136/jmg.2004.028712. PMID 15994879
- [Result] Govani FS, Shovlin CL. Fine mapping of the hereditary haemorrhagic telangiectasia (HHT)3 locus on chromosome 5 excludes VE-Cadherin-2, Sprouty4 and other interval genes. J Angiogenes Res. 2010 Aug 11;2:15. doi: 10.1186/2040-2384-2-15. PMID 20701797
- [Result] Clarke JM, Alikian M, Xiao S, Kasperaviciute D, Thomas E, Turbin I, Olupona K, Cifra E, Curetean E, Ferguson T, Redhead J; Genomics England Research Consortium; Shovlin CL. Low grade mosaicism in hereditary haemorrhagic telangiectasia identified by bidirectional whole genome sequencing reads through the 100,000 Genomes Project clinical diagnostic pipeline. J Med Genet. 2020 Dec;57(12):859-862. doi: 10.1136/jmedgenet-2019-106794. Epub 2020 Apr 17. No abstract available. PMID 32303606
- [Result] Shovlin CL, Simeoni I, Downes K, Frazer ZC, Megy K, Bernabeu-Herrero ME, Shurr A, Brimley J, Patel D, Kell L, Stephens J, Turbin IG, Aldred MA, Penkett CJ, Ouwehand WH, Jovine L, Turro E. Mutational and phenotypic characterization of hereditary hemorrhagic telangiectasia. Blood. 2020 Oct 22;136(17):1907-1918. doi: 10.1182/blood.2019004560. PMID 32573726
- [Result] Balachandar S, Graves TJ, Shimonty A, Kerr K, Kilner J, Xiao S, Slade R, Sroya M, Alikian M, Curetean E, Thomas E, McConnell VPM, McKee S, Boardman-Pretty F, Devereau A, Fowler TA, Caulfield MJ, Alton EW, Ferguson T, Redhead J, McKnight AJ, Thomas GA; Genomics England Research Consortium; Aldred MA, Shovlin CL. Identification and validation of a novel pathogenic variant in GDF2 (BMP9) responsible for hereditary hemorrhagic telangiectasia and pulmonary arteriovenous malformations. Am J Med Genet A. 2022 Mar;188(3):959-964. doi: 10.1002/ajmg.a.62584. Epub 2021 Dec 13. PMID 34904380
- [Result] Anderson E, Sharma L, Alsafi A, Shovlin CL. Pulmonary arteriovenous malformations may be the only clinical criterion present in genetically confirmed hereditary haemorrhagic telangiectasia. Thorax. 2022 Jun;77(6):628-630. doi: 10.1136/thoraxjnl-2021-218332. Epub 2022 Feb 14. PMID 35165143
- [Result] Joyce KE, Onabanjo E, Brownlow S, Nur F, Olupona K, Fakayode K, Sroya M, Thomas GA, Ferguson T, Redhead J, Millar CM, Cooper N, Layton DM, Boardman-Pretty F, Caulfield MJ; Genomics England Research Consortium; Shovlin CL. Whole genome sequences discriminate hereditary hemorrhagic telangiectasia phenotypes by non-HHT deleterious DNA variation. Blood Adv. 2022 Jul 12;6(13):3956-3969. doi: 10.1182/bloodadvances.2022007136. PMID 35316832
- [Result] Shovlin CL, Almaghlouth FI, Alsafi A, Coote N, Rennie C, Wallace GM, Govani FS, Research Consortium GE. Updates on diagnostic criteria for hereditary haemorrhagic telangiectasia in the light of whole genome sequencing of 'gene-negative' individuals recruited to the 100 000 Genomes Project. J Med Genet. 2024 Jan 19;61(2):182-185. doi: 10.1136/jmg-2023-109195. No abstract available. PMID 37586837
- [Result] Sharma L, Almaghlouth F, Mckernan H, Springett J, Tighe HC, Shovlin CL. Iron deficiency responses and integrated compensations in patients according to hereditary hemorrhagic telangiectasia ACVRL1, ENG and SMAD4 genotypes. Haematologica. 2024 Mar 1;109(3):958-962. doi: 10.3324/haematol.2022.282038. No abstract available. PMID 37731378